CLINICAL TRIAL: NCT06743178
Title: A Randomized Experiment to Test the Effects of Mass Media Photographs Related to Drug Use
Brief Title: The Effects of Mass Media Photographs on Drug-Related Stigma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Vital Strategies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00026173
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Opioid Use Disorder; Substance Use Disorders; Stigma, Social
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Social Stigma | interventions — Jails; Residence Characteristics; Salvage Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- No exposure control group (No Intervention): This group was not exposed to any drug-related photo.
- Photo of person injecting drugs (Experimental): Participants randomized to this arm were exposed to a photo of a person injecting drugs.
  Interventions: Behavioral: Photo of a person injecting drugs
- Photo of Emergency Medical Services (EMS) responding to an overdose (White) (Experimental): Participants randomized to this arm were exposed to a photo of EMS responding to a white person who had overdosed.
  Interventions: Behavioral: Photo of EMS responding to an overdose (White)
- Photo of EMS responding to an overdose (Black) (Experimental): Participants randomized to this arm were exposed to a photo of EMS responding to a Black person who had overdosed.
  Interventions: Behavioral: Photo of EMS responding to an overdose (Black)
- Photo of a person receiving treatment (Jail) (Experimental): Participants randomized to this arm were exposed to a photo of a person receiving methadone treatment in jail.
  Interventions: Behavioral: Photo of a person receiving treatment (Jail)
- Photo of a person receiving treatment (Community) (Experimental): Participants randomized to this arm were exposed to a photo of a person receiving methadone treatment in a community setting.
  Interventions: Behavioral: Photo of a person receiving treatment (Community)
- Photo of a person in recovery (White) (Experimental): Participants randomized to this arm were exposed to a photo of a white person in recovery in their workplace.
  Interventions: Behavioral: Photo of a person in recovery (White)
- Photo of a person in recovery (Black) (Experimental): Participants randomized to this arm were exposed to a photo of a Black person in recovery in their workplace.
  Interventions: Behavioral: Photo of a person in recovery (Black)
- Photo of a family member of an overdose decedent (Experimental): Participants randomized to this arm were exposed to a photo of a person who had lost a family member to an overdose.
  Interventions: Behavioral: Photo of a family member of an overdose decedent

INTERVENTIONS:
Behavioral: Photo of a person injecting drugs — Exposed to a photo of a person injecting drugs
  Arms: Photo of person injecting drugs
Behavioral: Photo of EMS responding to an overdose (White) — Exposed to a photo of EMS responding to an overdose (White)
  Arms: Photo of Emergency Medical Services (EMS) responding to an overdose (White)
Behavioral: Photo of EMS responding to an overdose (Black) — Exposed to a photo of EMS responding to an overdose (Black)
  Arms: Photo of EMS responding to an overdose (Black)
Behavioral: Photo of a person receiving treatment (Jail) — Exposed to a photo of a person receiving treatment (Jail)
  Arms: Photo of a person receiving treatment (Jail)
Behavioral: Photo of a person receiving treatment (Community) — Exposed to a photo of a person receiving treatment (Community)
  Arms: Photo of a person receiving treatment (Community)
Behavioral: Photo of a person in recovery (White) — Exposed to a photo of a person in recovery (White)
  Arms: Photo of a person in recovery (White)
Behavioral: Photo of a person in recovery (Black) — Exposed to a photo of a person in recovery (Black)
  Arms: Photo of a person in recovery (Black)
Behavioral: Photo of a family member of an overdose decedent — Exposed to a photo of a family member of an overdose decedent
  Arms: Photo of a family member of an overdose decedent

SUMMARY:
The aim of this study was to evaluate the effects of exposure to drug-related photos used by the media on emotions, stigma towards people who use drugs, and public health services for this population.

DETAILED DESCRIPTION:
This randomized experiment evaluated the impact of drug-related photographs used by the media on stigma towards people who use drugs. A nationally representative sample of US adults was randomized to view different photos used in the media (a person injecting drugs, a person being resuscitated after an overdose, a person receiving treatment, a person in recovery, or a person who had lost a family member to an overdose) and then asked questions about their feelings towards people who use drugs and their acceptance of public health services to address the overdose crisis.

ELIGIBILITY:
Inclusion Criteria:

* participant in existing web-based survey panel (NORC's AmeriSpeak)

Exclusion Criteria:

* not able to complete experiment and survey in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3570 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Affect Scale (Angry) | Immediately post-exposure to photo intervention
  Rating of feeling angry at the present moment. Item from the Positive and Negative Affect Scale. Measured on 5-point Likert scale with 1 indicating "not at all" and 5 indicating "extremely" their feeling angry at the present moment.
Positive and Negative Affect Scale (Sympathy) | Immediately post-exposure to photo intervention
  Rating of feeling sympathy at the present moment. Item from the Positive and Negative Affect Scale. Measured on 5-point Likert scale with 1 indicating "not at all" and 5 indicating "extremely" their feeling sympathy at the present moment.
Positive and Negative Affect Scale (Disgust) | Immediately post-exposure to photo intervention
  Rating of feeling disgust at the present moment. Item from the Positive and Negative Affect Scale. Measured on 5-point Likert scale with 1 indicating "not at all" and 5 indicating "extremely" their feeling disgust at the present moment.
Positive and Negative Affect Scale (Pity) | Immediately post-exposure to photo intervention
  Rating of feeling pity at the present moment. Item from the Positive and Negative Affect Scale. Measured on 5-point Likert scale with 1 indicating "not at all" and 5 indicating "extremely" their feeling pity at the present moment.
Social Distance Scale (Family) | Immediately post-exposure to photo intervention
  Rating of willingness to have person with substance use disorder marry into their family. Item from the Social Distance Scale that measures one element of stigma (desire for social distance). Measured on 5-point Likert scale with 1 indicating greater willingness and 5 indicating greater unwillingness to have a person with a substance use disorder marry into the family.
Social Distance Scale (Neighbor) | Immediately post-exposure to photo intervention
  Rating of willingness to have person with substance use disorder as a neighbor. Item from the Social Distance Scale that measures one element of stigma (desire for social distance). Measured on 5-point Likert scale with 1 indicating greater willingness and 5 indicating greater unwillingness to have a person with a substance use disorder as a neighbor.
Social Distance Scale (Work Closely) | Immediately post-exposure to photo intervention
  Rating of willingness to have person with substance use disorder work closely with them. Item from the Social Distance Scale that measures one element of stigma (desire for social distance). Measured on 5-point Likert scale with 1 indicating greater willingness and 5 indicating greater unwillingness to have a person with a substance use disorder work closely with them.
Social Distance Scale (close friend) | Immediately post-exposure to photo intervention
  Rating of willingness to have person with substance use disorder as a close personal friend. Item from the Social Distance Scale that measures one element of stigma (desire for social distance). Measured on 5-point Likert scale with 1 indicating greater willingness and 5 indicating greater unwillingness to have a person with a substance use disorder as a close personal friend.
Feeling-Thermometer measure of warmth towards people with substance use disorders | Immediately post-exposure to photo intervention
  Rating of warmth felt toward people with substance use disorder with 0 indicating extremely cold and 100 indicating extremely warm.
Rating of agreement that recovery is possible | Immediately post-exposure to photo intervention
  Rating of agreement with statement "Recovery from a drug addiction is possible" on a 5-point Likert scale with 1 indicating strongly agree and 5 indicating strongly disagree.
Rating of willingness to have a drug treatment program in their neighborhood | Immediately post-exposure to photo intervention
  Rating of willingness to have a drug treatment program in their neighborhood with 1 indicating greater willingness and 5 indicating greater unwillingness. Measured via survey questionnaire.
Rating of willingness to have a syringe exchange program in their neighborhood | Immediately post-exposure to photo intervention
  Rating of willingness to have a syringe exchange program in their neighborhood with 1 indicating greater willingness and 5 indicating greater unwillingness.
Rating of willingness to have a safe consumption site in their neighborhood | Immediately post-exposure to photo intervention
  Participant's rating of willingness to have a safe consumption site in their neighborhood with 1 indicating greater willingness and 5 indicating greater unwillingness.
Number of participants having a family member with a substance use disorder | Immediately post-exposure to photo intervention
  Personal experience of having a family member with a substance use disorder. Three close-ended response options (Yes, No, Don't know) when asked if the participant has ever had a family member with a substance use disorder.
Number of participants having a close friend with a substance use disorder | Immediately post-exposure to photo intervention
  Personal experience of having a close friend with a substance use disorder. Three close-ended response options (Yes, No, Don't know) when asked if the participant has ever had a close friend with a substance use disorder.
Number of participants having substance use disorder | Immediately post-exposure to photo intervention
  Personal experience of having a substance use disorder. Three close-ended response options (Yes; No; Don't Know) when asked if the participant has ever had a substance use disorder. Measured via survey questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Alene Kennedy-Hendricks, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hom JK, Heley K, Bandara S, Kennedy-Hendricks A. The impact of news photographs on drug-related stigma: A randomized message testing experiment in a National Sample of US Adults. Prev Med. 2025 Jun;195:108293. doi: 10.1016/j.ypmed.2025.108293. Epub 2025 Apr 29. PMID 40311941